CLINICAL TRIAL: NCT01662635
Title: CLINICOPATHOLOGICAL FEATURES OF NON-SMALL CELL LUNG CANCER PATIENTS ASSOCIATED WITH THE CHOROMOSOME 2p (EML4-ALK) INVERSION IN MEXICAN POPULATION.
Brief Title: Clinicopathological Features of NSCLC Patients Associated With the Chromosome 2p (EML4-ALK)
Acronym: ALK
Status: Completed | Type: Observational
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, MD and medical oncologist, Instituto Nacional de Cancerologia de Mexico
Other Study IDs: INCAN/CC/039/11
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2014-11-21 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2016-08

CONDITIONS: Non Small-cell Lung Cancer
Keywords: Non-small cell lung cancer.; Diagnosis,; Adenocarcinoma,; ALK,; FISH,; IHC; RT-qPCR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — FISH studies were performed in 3-mm to 4-mm thick paraffin sections from 230 NSCLCs and 1 ALCL specimen with t(2;5) that was used as a positive control for the break-apart detection.
  48 patients were analyzed for the presence of EML4-ALK gene fusion variants using the RNA from frozen tissue sections
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALK-BREAK APART: We reviewed 230 consecutive cases of NSCLC that were retrieved from oncologic molecular laboratory and diagnostic pathology unit at the Instituto Nacional de Cancerologia, Mexico city, between 2011 and 2014. Samples were sent to the unit of pathological anatomy, a Pathologist confirmed the histologic diagnosis. The only inclusion criterion was the availability of tissue for biomarker studies. Clinical and pathologic details of these patients were included in a database, obtained from medical records.
  For ALK fusion testing, we applied dual-color, break-apart FISH, RT-qPCR, and immunohistochemistry. Interpretation of the results was done in double-blind manner without knowing the results by other methods.

SUMMARY:
Because ALK-positive lung cancer constitutes less than 5% of all lung cancers, it is critically important to select those patients who are more likely to have the ALK mutation. Clinical characteristics of patients with mutations in the target gene should also be known, so that the incidence of a given target mutation is established in a specific population. There is not incidence known in Mexican population, but it is believed it is greater.

DETAILED DESCRIPTION:
Lung adenocarcinoma studies. The only inclusion criterion was the availability of tissue for biomarker studies. To identify ALK rearrangements, fluorescence in situ hybridization (FISH) studies were performed on 3 to 4 mm thick paraffin sections from NSCLCs. The commercially labeled Vysis LSI ALK Dual Color (split-apart), break-apart rearrangement probe (Abbott Molecular, Abbott Park, IL) was used to detect any rearrangement involving the ALK gene. The probe hybridizes to band 2p23, on either side of the ALK gene breakpoint. Criteria for probe signal interpretation in at least 200 interphase nuclei were as follow: 1) separated green and orange signals or single red signals identified cells with rearranged ALK; 2) overlapping of red and green signals (yellowish) indicated cells in which ALK was not rearranged.

FISH-positive samples for ALK rearrangement were defined as having cells with a clearly separated pair of probe signals, or with >15% of cells having loss of the 5´(centromeric) probe. The higher threshold for loss is necessary because parts of probes can be lost during sectioning.

The aim of our study is to evaluate the utility of IHC with 5A4 and RT-qPCR in the detection of ALK rearrangements in NSCLC compared with the current method of choice, FISH. Further, we report on the demographics, and clinicopathologic features of ALK-rearranged NSCLC in a Latin-American population.

Clinical details of these patients were included in a database. Further results will be analyzed with the program SPSS17

ELIGIBILITY:
Inclusion Criteria:

* The only inclusion criterion was the availability of tissue for biomarker studies.

Exclusion Criteria:

* Disease Progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mexican pupulation, with Non small-cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, Principal Investigator — Instituto de Cancerología
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jemal A, Freddie Bray, Melissa M, et al. Cancer statistics, 2011. CA Cancer J Clin. 61: 69-90, 2011. Wong DW. The EML4-ALK Fusion Gene Is Involved in Various Histologic Types of Lung Cancers From Non smokers With Wild-type EGFR and KRAS. Cancer 15, 1723-1733, 2009. Shaw, A. T. et al. Clinical Features and outcome of patients with non-small-cell lung cancer who harbor EML4-ALK. J. Clin. Oncol. 27, 4247-4253 2009. Kwak, E. L. et al. Anaplatic lymphoma kinase Inhibition in non-small cell lung cancer. N. Engl. J. Med. 363, 1693- 1703 2010. Soda M., Takada, S., Takeuchi, K., Choi, Y.L., Enomoto, M., Ueno, T. et al. A mouse model for EML4-ALK- positive lung cáncer. Proc Natl Acad Sci U S A 105: 19893-19897, 2008.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment began on February 01, 2011 and finished on September 01, 2014. All samples were obtained at the Instituto Nacional de Cancerología, in Mexico.
Pre-assignment Details: Samples were sent to the unit of Anatomic Pathology, where a pathologist confirmed the histologic diagnosis. The only inclusion criterion was the availability of tissue for biomarker studies.
Groups:
- Determination of ALK by FISH, IHC and RT-qPCR: The only inclusion criterion was the availability of tissue for biomarker studies.
  We use a commercially available break-apart probe kit specific to the ALK locus (Vysis LSI ALK Dual Color (split-apart); using the commercially mouse monoclonal ALK antibody for IHC and . Variants 1, 2, 3a, 4 and 5. The qPCR reactions were performed using the TaqMan Universal PCR MasterMix (Applied Biosystems/TaqMan, Life Technologies)
Period: Overall Study
Arm/Group | Determination of ALK by FISH, IHC and RT-qPCR
Started | 230
Completed | 200
Not Completed | 30
Not completed — scarce samples for evaluation | 30

BASELINE CHARACTERISTICS:
Population: The population evaluated included mexican patients, females and males, with ages between 18 and 80 years old, who had advanced lung cancer, who were referred to the Instituto Nacional de Cancerología in Mexico, between February 01, 2011 and September 01, 2014
Groups:
- Demographics and Clinical Features of Overall Population: The baseline characteristics of our population were on basis of the presence or absence of ALK gene.
Arm/Group | Demographics and Clinical Features of Overall Population
Number analyzed (Participants) | 200
Age, Customized [Number; unit: participants]
  < 55 years old | 91
  55 to 87 years old | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 87
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113
  Male | 87
Smoking history [Number; unit: participants]
  Non smokers ALK + | 12
  Smokers ALK+ | 7
  Non smokers ALK- | 95
  smokers ALK- | 86
ECOG Performance status [Number; unit: participants] — There were two groups:
  1. with an ECOG PS of 0-1( 0= Fully active, able to carry on all pre-disease performance without restriction, 1= Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work).
  2. ECOG PS of 2-3;( 2=Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours. 3=Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours).
  participants
    ECOG 0-1; ALK + | 15
    ECOG 2-3; ALK + | 4
    ECOG 0-1; ALK - | 148
    ECOG 2-3; ALK - | 33
Histology [Number; unit: participants]
  Squamus; ALK+ | 17
  Non-squamus; ALK + | 2
  Squamus; ALK - | 176
  Non-squamus; ALK - | 5
Wood smoke expossure [Number; unit: participants]
  Absent; ALK + | 9
  Present; ALK + | 10
  Absent; ALK - | 117
  Present; ALK - | 64
Histology Subtype [Number; unit: participants]
  Lepidic; ALK + | 3
  Acinar; ALK + | 5
  Papilar; ALK + | 2
  Micropapilar; ALK + | 1
  Solid; ALK + | 3
  Adenousquamous; ALK + | 0
  No otherwise specified; ALK + | 5
  Lepidic; ALK - | 14
  Acinar; ALK - | 39
  Papilar; ALK - | 13
  Micropapilar; ALK - | 10
  Solid; ALK - | 47
  Adenousquamous; ALK - | 16
  No otherwise specified; ALK - | 42

OUTCOME MEASURES:

1. Primary Outcome: FISH, IHC, RT-qPCR Comparison
Description: 200 samples underwent FISH, from them 63 underwent IHC and 48 RT-qPCR.
Time Frame: TWO YEARS
Population: The only selection criteria of our subjets was the availability of tumor tissue to perform tests.
Measure: Number; unit: participants
Groups:
- FISH Test: We use a commercially available break-apart probe kit specific to the ALK locus (Vysis LSI ALK Dual Color (split-apart); Abbott Molecular, Abbott Park, IL, USA). Slide washing, and counterstaining by DAPI were done following the manufacturer´s protocol (Abbott Molecular, Abbott Park, IL, USA).
- IHC Test: using the commercially mouse monoclonal ALK antibody (dilution 1:25, clone 5A4; Abcam, Cambridge, UK), with OptiView DAB detection Kit (Ventana, Tucson, Arizona, USA). ALK IHC was performed according to the protocols provided by the antibody.
- RT-qPCR Test: The qPCR reactions were performed using the TaqMan Universal PCR MasterMix (Applied Biosystems/TaqMan, Life Technologies) and the following Taqman assays: Hs03654556_ft (E13;A20), Hs03654557_ft (E20;A20), Hs03654558_ft (E6;A20), Hs03654560_ft (E17;A20), and Hs03654559_ft (E18;A20). Hs02758991_ft (GAPDH) assays, whose expression levels are known to be nearly stable among lung tumors
Arm/Group | FISH Test | IHC Test | RT-qPCR Test
Number analyzed (Participants) | 200 | 63 | 48
participants
  ALK+ | 18 | 15 | 5
  ALK- | 182 | 48 | 43
Statistical Analysis 1: Comparison: FISH Test vs IHC Test vs RT-qPCR Test; Continuous variables were summarized as arithmetic means, medians and standard deviations; and categorical variables were reported as proportions with 95% confidence intervals. Inferential comparisons were performed using Student's t test. The x2 or Fisher's exact tests were used to assess significance among categorical variables; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events not collected
Description: Adverse events not collected
Groups:
- Adverse Events Not Collected: "Serious and Other were not collected/assessed in this observational study."
Arm/Group | Adverse Events Not Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
There were no limitations in obtaining the planned number of samples. Two-hundred and thirty patients with advanced NSCLC were analyzed by FISH. Among the FISH tests performed, 30 were not evaluable due to scarce samples.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes